CLINICAL TRIAL: NCT05655832
Title: A Study to Investigate the Association of Real-world Sensor-derived Biometric Data With Clinical Parameters and Patient-reported Outcomes for Monitoring Disease Activity in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Study to Investigate the Association of Real-world Sensor-derived Biometric Data With Clinical Parameters and Patient-reported Outcomes for Monitoring Disease Activity in Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MS202559_0001
Record Dates: First submitted 2022-11-18; First posted 2022-12-19 (Actual); Results first posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COPD cohort (Experimental)
  Interventions: Device: Vivalink wearable device
- Calibration participants cohort (Experimental)
  Interventions: Device: Vivalink wearable device

INTERVENTIONS:
Device: Vivalink wearable device — a CE marked device modified to add a temperature measurement algorithm in addition to ECG and respiratory rate measurements

SUMMARY:
The purpose of this multicenter, prospective cohort study is to investigate the correlation of real-world sensor-derived biometric data obtained via a wearable device with clinical parameters and patient-reported outcomes (PROs) for monitoring disease activity and predicting exacerbations for participants with Chronic Obstructive Pulmonary Disease (COPD). The cohort of participants with COPD will be followed for 3 months. A calibration cohort with non-COPD participants will be included and followed for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

For participants with COPD:

* Participants ≥40 and ≤80 years at baseline
* Diagnosis of COPD stage II to IV
* History of moderate or severe exacerbations (≥2 moderate exacerbations or ≥1 severe exacerbations in any 12-month time window during last 3 years prior to inclusion and ≥1 moderate or severe exacerbations in the last 12 months prior to inclusion, considering that the last 12 months may reflect lower exacerbation rate due to Covid-19 measures)

For participants in the calibration cohort:

• Participants ≥40 and ≤80 years at baseline

Exclusion Criteria:

For participants with COPD:

* Clinically relevant and/or serious concurrent medical conditions including, but not limited to visual problems, severe mental illness or cognitive impairment, musculoskeletal or movement disorders, cardiac disease (e.g., heart failure, arrythmia [esp. atrial fibrillation and conduction blocks]), lung cancer (currently treated) that in the opinion of the Investigator, would interfere with participant's ability to participate in the study or draw meaningful conclusions from the study
* Participants with a cardiac pacemaker, defibrillators, or other implanted electronic devices
* Participants with known allergies or sensitivity to silicon or hydrogel
* Less than 6 weeks since previous moderate/severe exacerbation

For participants in the calibration cohort:

* Participants with a cardiac pacemaker, defibrillators, or other implanted electronic devices
* Participants with known allergies or sensitivity to silicon or hydrogel
* Diagnosis of pulmonary disease including, but not limited to COPD, asthma, pulmonary fibrosis, with impact on the lung function and exercise capacity

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (11):
- Germany (11):
  - Praxis an der Oper, Berlin
  - Lungenzentrum Darmstadt GmbH, Darmstadt
  - Städtische Kliniken Darmstadt, Darmstadt
  - Lungenzentrum Frankfurt, Frankfurt
  - Thoraxklinik Heidelberg gGmbH, Heidelberg
  - ZERO Praxen, Mannheim
  - Pneumologisches Studienzentrum München-West, München
  - Pneumologische Gemeinschaftspraxis Saarbrücken, Saarbrücken
  - RespiRatio / Lungenpraxis, Schleswig
  - Pneumologische Praxis Wiesbaden, Wiesbaden
  - Lungenpraxis Dr. Franz / Dr. Weber, Witten

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website http://bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS202559_0001

RESULTS

PARTICIPANT FLOW:
Groups:
- Calibration Cohort: Participants in this group did not have COPD and wore a Vivalink wearable device and were observed for a period of 2 weeks
- COPD Cohort: Participants in this group wore a Vivalink wearable device and were observed for a period of 3 months.
Period: Overall Study
Arm/Group | Calibration Cohort | COPD Cohort
Started | 10 | 67
Completed | 10 | 64
Not Completed | 0 | 3
Not completed — Not mentioned | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol non-compliance | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intention-To-Treat (ITT) population consisted of the following analysis sets: COPD analysis set: all eligible participants with COPD & Calibration analysis set: all eligible participants with non-COPD
Groups:
- Total: Total of all reporting groups
Arm/Group | Calibration Cohort | COPD Cohort | Total
Number analyzed (Participants) | 10 | 67 | 77
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 52 [43.75 to 58.75] | 67 [61 to 71.5] | 66 [59 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 37 | 45
  Male | 2 | 30 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 67 | 77
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Chronic Obstructive Pulmonary Disease (COPD) Exacerbations of Sensor-collected Parameters During Observation Period - Physical Activity
Description: An activity flag is extracted from the accelerometer by Vivalink, by using a predefined threshold for adult movement. For stair climbing, first periodic movement was determined, by using frequency analysis on specific time windows, and generating a ratio to the total spectrum indicating periodic activity over a certain threshold.
Time Frame: Day 0(Baseline) and Day 8 to Day 14
Population: COPD cohort consisted of all participants with COPD fulfilling all of the inclusion criteria and none of the exclusion criteria. Here, "Number analyzed" signifies those participants who were evaluable at specified time point
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | COPD Cohort
Number analyzed (Participants) | 67
minutes
  Day 0: number analyzed (Participants) | 62
  Day 0 | 41.98 (22.89)
  Day 8 to Day 14 | 58.93 (33.026)

2. Primary Outcome: Chronic Obstructive Pulmonary Disease (COPD) Exacerbations of Sensor-collected Parameters During Observation Period - Heart Rate
Description: Heart rate is provided by Vivalink.
Time Frame: Day 0(Baseline) and Day 8 to Day 14
Population: COPD cohort consists of all participants with COPD fulfilling all of the inclusion criteria and none of the exclusion criteria. Here, "Number analyzed" signifies those participants who were evaluable at specified time point.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | COPD Cohort
Number analyzed (Participants) | 67
beats per minute
  Day 0: number analyzed (Participants) | 62
  Day 0 | 86.4 (7.953)
  Day 8 to Day 14 | 81.26 (9.237)

3. Primary Outcome: Chronic Obstructive Pulmonary Disease (COPD) Exacerbations of Sensor-collected Parameters During Observation Period - Heart Rate Variability (SDRR, SDNN, SDNNI, RMSSD, ln(RMSSD))
Description: Heart rate variability reflecting differences in time intervals between 2 R-waves in the ECG (milliseconds) SDRR (Standard Deviation of Intervals between Heartbeats), SDNN (Standard Deviation of Intervals between Heartbeats, after removing abnormal Beats), SDNNI (Mean of the Standard Deviations of all the NN intervals for each 5 min Segment of a 24-h HRV Recording), and RMSSD (Mean of the Standard Deviations of all the NN intervals for each 5 min Segment of a 24-hour HRV Recording) and In(RMSDD)
Time Frame: Day 0(Baseline) and Day 8 to Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | COPD Cohort
Number analyzed (Participants) | 67
milliseconds
  SDRR: Day 0: number analyzed (Participants) | 61
  SDRR: Day 0 | 26.83 (11.37)
  SDRR: Day 8-14 | 23.34 (10.867)
  SDNN: Day 0: number analyzed (Participants) | 61
  SDNN: Day 0 | 58.71 (47.79)
  SDNN: Day 8-14 | 52.82 (39.419)
  SDNNI: Day 0: number analyzed (Participants) | 61
  SDNNI: Day 0 | 69.51 (63.18)
  SDNNI: Day 8-14 | 63.18 (33.537)
  RMSSD: Day 0: number analyzed (Participants) | 61
  RMSSD: Day 0 | 55.37 (59.658)
  RMSSD: Day 8-14 | 53.73 (73.024)
  In (RMSSD): Day 0: number analyzed (Participants) | 61
  In (RMSSD): Day 0 | 3.59 (0.883)
  In (RMSSD): Day 8-14 | 3.51 (0.813)

4. Primary Outcome: Chronic Obstructive Pulmonary Disease (COPD) Exacerbations of Sensor-collected Parameters During Observation Period - Heart Rate Variability (pNN50)
Description: pNN50 is the percentage of adjacent NN intervals that differ from each other by more than 50 milliseconds.
Time Frame: Day 0(Baseline) and Day 8 to Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | COPD Cohort
Number analyzed (Participants) | 67
percentage
  Day 0: number analyzed (Participants) | 61
  Day 0 | 0.12 (0.198)
  Day 8-14 | 0.11 (0.197)

5. Primary Outcome: Chronic Obstructive Pulmonary Disease (COPD) Exacerbations of Sensor-collected Parameters During Observation Period - Heart Rate Variability (Stress Index)
Description: Baevsky's Stress Index is a heart rate variability (HRV) measure used to assess autonomic nervous system activity and physiological stress, especially in monitoring chronic obstructive pulmonary disease (COPD) exacerbations. It is calculated as: amplitude of the mode (AMo) divided by two times the mode (Mo) multiplied by the difference between the maximum and minimum RR intervals (MxDMn). AMo is the percentage of RR intervals at the most frequent value, Mo is the most common RR interval, and MxDMn is the range of RR intervals. The index typically ranges from 50 to over 900. Lower values (50-150) indicate low stress and better autonomic balance, while higher values (above 500) reflect increased stress and sympathetic activity. Values above 900 are considered very high stress. This is a single composite score with no subscales; higher scores represent worse outcomes.
Time Frame: Day 0(Baseline) and Day 8 to Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | COPD Cohort
Number analyzed (Participants) | 67
ratio
  Day 0: number analyzed (Participants) | 61
  Day 0 | 108.43 (94.236)
  Day 8-14 | 99.86 (81.076)

6. Primary Outcome: Chronic Obstructive Pulmonary Disease (COPD) Exacerbations of Sensor-collected Parameters During Observation Period - Heart Rate Variability (LF and HF)
Description: Applying a Fast Fourier Transformation (FFT) or autoregressive (AR) modeling one can separate Heart rate variability (HRV) into its component ultra-low-frequency (ULF), very low frequency (VLF), Low-Frequency power (LF), and High-Frequency power (HF) rhythms that operate within different frequency ranges. Given in absolute values of power (milliseconds squared). LF power, low frequency power (0.04-0.15 Hz). HF power, high frequency power (0.15-0.40 Hz). LF/HF Ratio, spectral HRV index computed as (LF/HF).
Time Frame: Day 0(Baseline) and Day 8 to Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hertz
Arm/Group | COPD Cohort
Number analyzed (Participants) | 67
hertz
  LF: Day 0: number analyzed (Participants) | 61
  LF: Day 0 | 320.32 (456.411)
  LF: Day 8-14 | 287.19 (399.897)
  HF: Day 0: number analyzed (Participants) | 61
  HF: Day 0 | 646.3 (1234.891)
  HF: Day 8-14 | 612.6 (1542.947)

7. Primary Outcome: Chronic Obstructive Pulmonary Disease (COPD) Exacerbations of Sensor-collected Parameters During Observation Period - Heart Rate Variability (LF/HF)
Description: as for outcome 6
Time Frame: Day 0(Baseline) and Day 8 to Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | COPD Cohort
Number analyzed (Participants) | 67
ratio
  LF/HF: Day 0: number analyzed (Participants) | 61
  LF/HF: Day 0 | 1.38 (1.211)
  LF/HF: Day 8-14 | 1.51 (1.204)

8. Primary Outcome: Chronic Obstructive Pulmonary Disease (COPD) Exacerbations of Sensor-collected Parameters During Observation Period - Temperature
Description: Temperature is provided by Vivalink. The value for temperature is derived by Vivalink from the display temperature and then calibrated using initial calibration values, in an IP protected process. The sensor temperature is considered only as a relative value to evaluate changes in the temperature, and not as an objective human body temperature value, meaning no thresholds relative to normal human body temperature are considered, and it will not be used as a marker for fever or hypothermia.
Time Frame: Day 0(Baseline) and Day 8 to Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: celsius
Arm/Group | COPD Cohort
Number analyzed (Participants) | 67
celsius
  Day 0: number analyzed (Participants) | 62
  Day 0 | 36.77 (1.155)
  Day 8 to 14 | 37.14 (1.239)

9. Primary Outcome: Chronic Obstructive Pulmonary Disease (COPD) Exacerbations of Sensor-collected Parameters During Observation Period - Respiratory Rate
Description: Respiration rate is provided by Vivalink.
Time Frame: Day 0(Baseline) and Day 8 to Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | COPD Cohort
Number analyzed (Participants) | 67
breaths per minute
  Day 0: number analyzed (Participants) | 62
  Day 0 | 21.42 (1.903)
  Day 8 to Day 14 | 20.92 (2.247)

10. Primary Outcome: Chronic Obstructive Pulmonary Disease (COPD) Exacerbations of Sensor-collected Parameters During Observation Period - Cough Frequency
Description: Cough Frequency was provided by vivalink.
Time Frame: Day 0(Baseline) and Day 8 to Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: count per day
Arm/Group | COPD Cohort
Number analyzed (Participants) | 67
count per day
  Day 0: number analyzed (Participants) | 62
  Day 0 | 56.82 (48.46)
  Day 8 to Day 14 | 72.46 (58.62)

11. Primary Outcome: Chronic Obstructive Pulmonary Disease (COPD) Exacerbations of Sensor-collected Parameters During Observation Period - Sleep Patterns
Description: The basis of the sleep pattern calculations is the self-reported bedtimes. With the same technique as the cough frequency prediction, inactivity signals can be predicted from the labeled data to improve the bedtime accuracy, and the changes in accelerometer (step detection algorithms) can be used to quantify the number of clear breaks in the sleep (standing up, strong cough, etc.).
Time Frame: Day 0(Baseline) and Day 8 to Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | COPD Cohort
Number analyzed (Participants) | 67
hours
  Day 0: number analyzed (Participants) | 62
  Day 0 | 8.7 (1.892)
  Day 8 to Day 14: number analyzed (Participants) | 66
  Day 8 to Day 14 | 8.48 (1.491)

12. Primary Outcome: Chronic Obstructive Pulmonary Disease (COPD) Exacerbations of Sensor-collected Parameters During Observation Period - Resting Heart Rate
Description: Resting Heart Rate is provided by Vivalink.
Time Frame: Day 0(Baseline) and Day 8 to Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | COPD Cohort
Number analyzed (Participants) | 67
beats per minute
  Day 0: number analyzed (Participants) | 62
  Day 0 | 85.02 (8.003)
  Day 8 to Day 14 | 79.9 (9.126)

13. Primary Outcome: Chronic Obstructive Pulmonary Disease (COPD) Exacerbations of Sensor-collected Parameters During Observation Period - Inspiration vs Expiration Time Ratio
Description: Using the breathing signal one can determine the inspiration and expiration peaks. The difference between said peaks in milliseconds can be used to determine the ratio of inspiration (distance from lower point to next peak) vs expiration (distance from peak to next lower point).
Time Frame: Day 0(Baseline) and Day 8 to Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | COPD Cohort
Number analyzed (Participants) | 67
ratio
  Day 0: number analyzed (Participants) | 61
  Day 0 | 0.96 (0.078)
  Day 8 to Day 14 | 0.98 (0.068)

14. Primary Outcome: Chronic Obstructive Pulmonary Disease (COPD) Exacerbations of Sensor-collected Parameters During Observation Period - Frequency of Additional Medication
Description: Count of the number of times the use of additional medication as a log activity is reported per day.
Time Frame: Day 0(Basseline) and Day 8 to Day 14
Population: COPD cohort consisted of all participants with COPD fulfilling all of the inclusion criteria and none of the exclusion criteria.
Measure: Mean (Standard Deviation); unit: count per day
Arm/Group | COPD Cohort
Number analyzed (Participants) | 67
count per day
  Day 0 | 0.37 (0.714)
  Day 8 to Day 14 | 0.82 (0.859)

15. Primary Outcome: Prediction of Moderate or Severe COPD Exacerbations by Building a Statistical Model Employing Sensor-Derived Data and Demographic and Medical Covariates - Accuracy
Description: Accuracy was calculated as (True Positives + True Negatives) / Total Population. True Positives (TP) are events correctly predicted as exacerbations. True Negatives (TN) are events correctly predicted as non-exacerbations. Total Population refers to the total number of events evaluated. Accuracy scores reflect XGBoost algorithm performance using random and time-based 70/30 data splits. The values were calculated in form of percentage where 100% is the ideal scenario for perfect predictability.
Time Frame: Up to 3 months
Population: as for outcome 14
Measure: Number; unit: percentage of predictability
Arm/Group | COPD Cohort
Number analyzed (Participants) | 67
percentage of predictability
  70-30 | 0.56
  Random | 0.56

16. Primary Outcome: Prediction of Moderate or Severe COPD Exacerbations by Building a Statistical Model Employing Sensor-Derived Data and Demographic and Medical Covariates - Precision
Description: Precision was calculated as True Positives / (True Positives + False Positives). True Positives (TP) are events correctly predicted as exacerbations. False Positives (FP) are events incorrectly predicted as exacerbations. Total Population refers to the total number of events evaluated. Precision scores reflect XGBoost algorithm performance using random and time-based 70/30 data splits. The values were calculated in form of percentage where 100% is the ideal scenario for perfect predictability.
Time Frame: Up to 3 months
Population: as for outcome 14
Measure: Number; unit: percentage of predictability
Arm/Group | COPD Cohort
Number analyzed (Participants) | 67
percentage of predictability
  70-30 | 0.53
  Random | 0.62

17. Primary Outcome: Prediction of Moderate or Severe COPD Exacerbations by Building a Statistical Model Employing Sensor-Derived Data and Demographic and Medical Covariates - Recall
Description: Recall was calculated as True Positives / (True Positives + False Negatives). True Positives (TP) are events correctly predicted as exacerbations. False Negatives (FN) are events incorrectly predicted as non-exacerbations. Total Population refers to the total number of events evaluated. Recall scores reflect XGBoost algorithm performance using random and time-based 70/30 data splits. The values were calculated in form of percentage where 100% is the ideal scenario for perfect predictability.
Time Frame: Up to 3 months
Population: as for outcome 14
Measure: Number; unit: percentage of predictability
Arm/Group | COPD Cohort
Number analyzed (Participants) | 67
percentage of predictability
  70-30 | 0.63
  Random | 0.46

18. Primary Outcome: Prediction of Moderate or Severe COPD Exacerbations by Building a Statistical Model Employing Sensor-Derived Data and Demographic and Medical Covariates - Specificity
Description: Specificity was calculated as True Negatives / (True Negatives + False Positives). True Negatives (TN) are events correctly predicted as non-exacerbations. False Positives (FP) are events incorrectly predicted as exacerbations. Total Population refers to the total number of events evaluated. Specificity scores reflect XGBoost algorithm performance using random and time-based 70/30 data splits. The values were calculated in form of percentage where 100% is the ideal scenario for perfect predictability.
Time Frame: Up to 3 months
Population: as for outcome 14
Measure: Number; unit: percentage of predictability
Arm/Group | COPD Cohort
Number analyzed (Participants) | 67
percentage of predictability
  70-30 | 0.53
  Random | 0.63

19. Secondary Outcome: Correlation of Sensor-Collected Data With COPD Assessment Test (CAT) Questionnaire: Participants Health Status and Symptoms at Baseline and Study End
Description: Participants health status and symptoms at baseline (Day 0) and study end will be measured as the summary score across items of the CAT questionnaire that consists of 8-items in which participants can choose a score from 0 to 5, for each visit.
Time Frame: Baseline (Day 0) and at 3 months
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | COPD Cohort
Number analyzed (Participants) | 67
correlation coefficient
  Baseline: Heart Rate | 0.19 [-0.07 to 0.43]
  End of Study: Heart Rate | 0.45 [0.16 to 1.67]
  Baseline: Resting Heart Rate | 0.19 [-0.07 to 0.43]
  End of Study: Resting Heart Rate | 0.46 [0.16 to 0.68]
  Baseline: Temperature | 0.07 [-0.19 to 0.32]
  End of Study: Temperature | 0.02 [-0.31 to 0.33]
  Baseline: Temperature (normalized) | 0.12 [-0.14 to 0.36]
  End of Study: Temperature (normalized) | -0.13 [-0.43 to 0.2]
  Baseline: Respiration Rate | 0.21 [-0.05 to 0.44]
  End of Study: Respiration Rate | 0.3 [-0.02 to 0.57]
  Baseline: SDRR | 0.04 [-0.22 to 0.3]
  End of Study: SDRR | 0.39 [0.08 to 0.63]
  Baseline: SDNN | -0.06 [-0.31 to 0.21]
  End of Study: SDNN | 0.38 [0.07 to 0.63]
  Baseline: SDNNI | 0.02 [-0.24 to 0.28]
  End of Study: SDNNI | 0.41 [0.09 to 0.65]
  Baseline: RMSSD | -0.04 [-0.29 to 0.22]
  End of Study: RMSSD | 0.42 [0.12 to 0.66]
  Baseline: In (RMSSD) | 0.04 [-0.22 to 0.29]
  End of Study: In (RMSSD) | 0.44 [0.14 to 0.67]
  Baseline: pNN50 | -0.06 [-0.31 to 0.2]
  End of Study: pNN50 | 0.4 [0.09 to 0.64]
  Baseline: Stress Index | -0.01 [-0.27 to 0.25]
  End of Study: Stress Index | -0.21 [-0.5 to 0.12]
  Baseline: LF | -0.28 [-0.5 to -0.03]
  End of Study: LF | 0.15 [-0.19 to 0.45]
  Baseline: HF | -0.09 [-0.34 to 0.17]
  End of Study: HF | 0.18 [-0.16 to 0.47]
  Baseline: LF/HF | -0.12 [-0.36 to 0.15]
  End of Study: LF/ HF | -0.34 [-0.6 to -0.01]
  Baseline: Physical Activity | -0.11 [-0.36 to 0.15]
  End of Study: Physical Activity | -0.11 [-0.42 to 0.22]
  Baseline: Physical Activity (normalized) | 0.06 [-0.2 to 0.31]
  End of Study: Physical Activity (normalized) | 0.11 [-0.22 to 0.42]
  Baseline: In- vs. Expiration Time Ratio | -0.04 [-0.3 to 0.22]
  End of Study: In- vs. Expiration Time Ratio | -0.21 [-0.5 to 0.12]
  Baseline: Cough Frequency | -0.2 [-0.43 to 0.06]
  End of Study: Cough Frequency | -0.21 [-0.5 to 0.12]
  Baseline: Cough Frequency (normalized) | 0.06 [-0.2 to 0.31]
  End of Study: Cough Frequency (normalized) | 0.27 [-0.06 to 0.55]

20. Secondary Outcome: Correlation of Sensor-Collected Data With Lung Function (FEV1) at Baseline and Study End
Description: Lung function was assessed using plethysmography.
Time Frame: Baseline (Day 0) and at 3 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | COPD Cohort
Number analyzed (Participants) | 39
correlation coefficient
  Baseline: Heart Rate | 0.07 [-0.23 to 0.35]
  End of Study: Heart Rate | -0.36 [-0.62 to -0.01]
  Baseline: Resting Heart Rate | 0.08 [-0.22 to 0.36]
  End of Study: Resting Heart Rate | -0.32 [-0.6 to 0.03]
  Baseline: Temperature | -0.29 [-0.54 to -0.01]
  End of Study: Temperature | -0.12 [-0.45 to 0.23]
  Baseline: Temperature (normalized) | -0.18 [-0.45 to 0.11]
  End of Study: Temperature (normalized) | 0.1 [-0.25 to 0.43]
  Baseline: Respiration Rate | -0.25 [-0.5 to 0.04]
  End of Study: Respiration Rate | -0.24 [-0.54 to 0.11]
  Baseline: SDRR | -0.28 [-0.53 to 0.01]
  End of Study: SDRR | -0.31 [-0.6 to 0.04]
  Baseline: SDNN | 0.15 [-0.14 to 0.42]
  End of Study: SDNN | -0.17 [-0.49 to 0.19]
  Baseline: SDNNI | -0.02 [-0.31 to 0.27]
  End of Study: SDNNI | -0.25 [-0.55 to 0.11]
  Baseline: RMSSD | 0.08 [-0.21 to 0.36]
  End of Study: RMSSD | -0.19 [-0.5 to 0.17]
  Baseline: In (RMSSD) | 0.02 [-0.27 to 0.3]
  End of Study: In (RMSSD) | -0.17 [-0.49 to 0.19]
  Baseline: pNN50 | 0.05 [-0.24 to 0.33]
  End of Study: pNN50 | -0.16 [-0.48 to 0.2]
  Baseline: Stress Index | -0.04 [-0.32 to 0.25]
  End of Study: Stress Index | -0.09 [-0.42 to 0.27]
  Baseline: LF | 0.35 [0.07 to 0.58]
  End of Study: LF | -0.11 [-0.44 to 0.25]
  Baseline: HF | 0.18 [-0.11 to 0.45]
  End of Study: HF | -0.14 [-0.46 to 0.22]
  Baseline: LF/HF | 0.14 [-0.15 to 0.41]
  End of Study: LF/ HF | 0.04 [-0.32 to 0.38]
  Baseline: Physical Activity | 0.11 [-0.18 to 0.39]
  End of Study: Physical Activity | -0.03 [-0.37 to 0.32]
  Baseline: Physical Activity (normalized) | -0.09 [-0.37 to 0.2]
  End of Study: Physical Activity (normalized) | -0.24 [-0.54 to 0.11]
  Baseline: In- vs. Expiration Time Ratio | 0.29 [0 to 0.53]
  End of Study: In- vs. Expiration Time Ratio | 0.13 [-0.23 to 0.46]
  Baseline: Cough Frequency | 0.18 [-0.11 to 0.45]
  End of Study: Cough Frequency | -0.05 [-0.39 to 0.3]
  Baseline: Cough Frequency (normalized) | 0.02 [-0.27 to 0.3]
  End of Study: Cough Frequency (normalized) | -0.2 [-0.51 to 0.15]

21. Secondary Outcome: Correlation of Sensor-Collected Data With Lung Function (FVC) at Baseline and Study End
Description: Lung function was assessed using plethysmography.
Time Frame: Baseline (Day 0) and at 3 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | COPD Cohort
Number analyzed (Participants) | 39
correlation coefficient
  Baseline: Heart Rate | 0.11 [-0.18 to 0.38]
  End of Study: Heart Rate | -0.15 [-0.47 to 0.21]
  Baseline: Resting Heart Rate | 0.13 [-0.16 to 0.4]
  End of Study: Resting Heart Rate | -0.11 [-0.44 to 0.24]
  Baseline: Temperature | -0.21 [-0.47 to 0.08]
  End of Study: Temperature | -0.28 [-0.57 to 0.07]
  Baseline: Temperature (normalized) | -0.32 [-0.55 to -0.03]
  End of Study: Temperature (normalized) | -0.1 [-0.43 to 0.25]
  Baseline: Respiration Rate | -0.28 [-0.52 to 0.01]
  End of Study: Respiration Rate | -0.09 [-0.42 to 0.26]
  Baseline: SDRR | -0.2 [-0.46 to 0.09]
  End of Study: SDRR | -0.04 [-0.38 to 0.31]
  Baseline: SDNN | 0.16 [-0.13 to 0.43]
  End of Study: SDNN | 0.09 [-0.27 to 0.43]
  Baseline: SDNNI | 0.03 [-0.26 to 0.31]
  End of Study: SDNNI | 0.04 [-0.31 to 0.38]
  Baseline: RMSSD | 0.1 [-0.19 to 0.38]
  End of Study: RMSSD | 0.19 [-0.17 to 0.5]
  Baseline: In (RMSSD) | 0.04 [-0.25 to 0.32]
  End of Study: In (RMSSD) | 0.03 [-0.32 to 0.38]
  Baseline: pNN50 | 0.07 [-0.22 to 0.35]
  End of Study: pNN50 | 0.21 [-0.15 to 0.52]
  Baseline: Stress Index | -0.09 [-0.36 to 0.21]
  End of Study: Stress Index | 0.25 [-0.11 to 0.55]
  Baseline: LF | 0.31 [0.02 to 0.55]
  End of Study: LF | 0.29 [-0.06 to 0.58]
  Baseline: HF | 0.15 [-0.14 to 0.42]
  End of Study: HF | 0.32 [-0.04 to 0.6]
  Baseline: LF/HF | 0.25 [-0.04 to 0.5]
  End of Study: LF/ HF | 0.04 [-0.32 to 0.38]
  Baseline: Physical Activity | 0.02 [-0.27 to 0.3]
  End of Study: Physical Activity | 0.11 [-0.24 to 0.44]
  Baseline: Physical Activity (normalized) | -0.07 [-0.35 to 0.22]
  End of Study: Physical Activity (normalized) | 0.09 [-0.26 to 0.42]
  Baseline: In- vs. Expiration Time Ratio | 0.22 [-0.07 to 0.48]
  End of Study: In- vs. Expiration Time Ratio | 0.02 [-0.33 to 0.36]
  Baseline: Cough Frequency | 0.16 [-0.13 to 0.43]
  End of Study: Cough Frequency | -0.16 [-0.47 to 0.2]
  Baseline: Cough Frequency (normalized) | 0.12 [-0.17 to 0.4]
  End of Study: Cough Frequency (normalized) | 0.06 [-0.28 to 0.4]

22. Secondary Outcome: Correlation of Sensor-Collected Data With Lung Function (FEV1/FVC) at Baseline and Study End
Description: Lung function was assessed using plethysmography.
Time Frame: Baseline (Day 0) and at 3 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | COPD Cohort
Number analyzed (Participants) | 39
correlation coefficient
  Baseline: Heart Rate | -0.07 [-0.35 to 0.22]
  End of Study: Heart Rate | -0.3 [-0.59 to 0.04]
  Baseline: Resting Heart Rate | -0.08 [-0.36 to 0.21]
  End of Study: Resting Heart Rate | -0.29 [-0.58 to 0.05]
  Baseline: Temperature | -0.16 [-0.43 to 0.14]
  End of Study: Temperature | 0.15 [-0.2 to 0.47]
  Baseline: Temperature (normalized) | 0.07 [-0.22 to 0.35]
  End of Study: Temperature (normalized) | 0.28 [-0.07 to 0.57]
  Baseline: Respiration Rate | 0 [-0.29 to 0.28]
  End of Study: Respiration Rate | -0.22 [-0.52 to 0.14]
  Baseline: SDRR | -0.27 [-0.51 to 0.02]
  End of Study: SDRR | -0.42 [-0.67 to -0.08]
  Baseline: SDNN | -0.08 [-0.36 to 0.21]
  End of Study: SDNN | -0.28 [-0.57 to 0.08]
  Baseline: SDNNI | -0.17 [-0.44 to 0.12]
  End of Study: SDNNI | -0.35 [-0.63 to -0.01]
  Baseline: RMSSD | -0.09 [-0.37 to 0.2]
  End of Study: RMSSD | -0.36 [-0.63 to -0.01]
  Baseline: In (RMSSD) | -0.13 [-0.4 to 0.16]
  End of Study: In (RMSSD) | -0.23 [-0.53 to 0.13]
  Baseline: pNN50 | -0.09 [-0.37 to 0.2]
  End of Study: pNN50 | -0.33 [-0.61 to 0.02]
  Baseline: Stress Index | 0.09 [-0.2 to 0.37]
  End of Study: Stress Index | -0.31 [-0.59 to 0.05]
  Baseline: LF | 0.07 [-0.22 to 0.35]
  End of Study: LF | -0.31 [-0.59 to 0.05]
  Baseline: HF | 0.02 [-0.27 to 0.31]
  End of Study: HF | -0.36 [-0.63 to -0.01]
  Baseline: LF/HF | -0.06 [-0.34 to 0.23]
  End of Study: LF/ HF | 0.03 [-0.33 to 0.37]
  Baseline: Physical Activity | 0.2 [-0.09 to 0.46]
  End of Study: Physical Activity | -0.15 [-0.47 to 0.2]
  Baseline: Physical Activity (normalized) | -0.02 [-0.31 to 0.26]
  End of Study: Physical Activity (normalized) | -0.37 [-0.64 to -0.03]
  Baseline: In- vs. Expiration Time Ratio | 0.2 [-0.09 to 0.46]
  End of Study: In- vs. Expiration Time Ratio | 0.17 [-0.19 to 0.49]
  Baseline: Cough Frequency | -0.02 [-0.31 to 0.27]
  End of Study: Cough Frequency | 0.1 [-0.25 to 0.43]
  Baseline: Cough Frequency (normalized) | -0.18 [-0.44 to 0.12]
  End of Study: Cough Frequency (normalized) | -0.29 [-0.57 to 0.06]

23. Secondary Outcome: Correlation of Sensor-Collected Data With COPD Assessment Test (CAT) Questionnaire: Lung Function and Lab Values at Baseline and Study End (White Blood Cells Count)
Description: Lung function was assessed using plethysmography and lab values including Complete Blood Count with differential, Blood Gas Analysis, procalcitonin and CRP will be assessed as per standard practice at baseline (Day 0) and at study end
Time Frame: Baseline (Day 0) and at 3 months
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | COPD Cohort
Number analyzed (Participants) | 67
correlation coefficient
  Baseline: Heart Rate | 0.2 [-0.25 to 0.58]
  End of Study: Heart Rate | -0.07 [-0.5 to 0.39]
  Baseline: Resting Heart Rate | 0.21 [-0.24 to 0.59]
  End of Study: Resting Heart Rate | -0.04 [-0.47 to 0.41]
  Baseline: Temperature | 0.19 [-0.26 to 0.58]
  End of Study: Temperature | 0.34 [-0.12 to 0.68]
  Baseline: Temperature (normalized) | -0.29 [-0.64 to 0.16]
  End of Study: Temperature (normalized) | 0.38 [-0.08 to 0.7]
  Baseline: Respiration Rate | 0.42 [-0.02 to 0.72]
  End of Study: Respiration Rate | -0.06 [-0.49 to 0.4]
  Baseline: SDRR | 0.12 [-0.33 to 0.53]
  End of Study: SDRR | -0.01 [-0.46 to 0.44]
  Baseline: SDNN | 0.22 [-0.24 to 0.59]
  End of Study: SDNN | 0.21 [-0.27 to 0.61]
  Baseline: SDNNI | 0.28 [-0.17 to 0.63]
  End of Study: SDNNI | 0.12 [-0.35 to 0.55]
  Baseline: RMSSD | 0.31 [-0.14 to 0.65]
  End of Study: RMSSD | 0.25 [-0.23 to 0.63]
  Baseline: In (RMSSD) | 0.25 [-0.2 to 0.62]
  End of Study: In (RMSSD) | 0.32 [-0.16 to 0.68]
  Baseline: pNN50 | 0.4 [-0.04 to 0.71]
  End of Study: pNN50 | 0.34 [-0.14 to 0.69]
  Baseline: Stress Index | 0.02 [-0.42 to 0.45]
  End of Study: Stress Index | -0.23 [-0.62 to 0.25]
  Baseline: LF | -0.1 [-0.51 to 0.35]
  End of Study: LF | 0.37 [-0.1 to 0.71]
  Baseline: HF | -0.1 [-0.51 to 0.35]
  End of Study: HF | 0.42 [-0.04 to 0.74]
  Baseline: LF/HF | -0.07 [-0.49 to 0.37]
  End of Study: LF/ HF | -0.3 [-0.66 to 0.18]
  Baseline: Physical Activity | -0.41 [-0.72 to 0.02]
  End of Study: Physical Activity | -0.19 [-0.59 to 0.27]
  Baseline: Physical Activity (normalized) | -0.36 [-0.68 to 0.09]
  End of Study: Physical Activity (normalized) | 0.13 [-0.33 to 0.54]
  Baseline: In- vs. Expiration Time Ratio | -0.17 [-0.56 to 0.28]
  End of Study: In- vs. Expiration Time Ratio | -0.05 [-0.49 to 0.41]
  Baseline: Cough Frequency | 0.02 [-0.41 to 0.45]
  End of Study: Cough Frequency | 0.26 [-0.21 to 0.63]
  Baseline: Cough Frequency (normalized) | -0.27 [-0.63 to 0.19]
  End of Study: Cough Frequency (normalized) | -0.31 [-0.66 to 0.15]

24. Secondary Outcome: Correlation of Sensor-Collected Data With COPD Assessment Test (CAT) Questionnaire: Lung Function and Lab Values at Baseline and Study End (Erythrocytes Count)
Description: as for outcome 23
Time Frame: Baseline (Day 0) and at 3 months
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | COPD Cohort
Number analyzed (Participants) | 67
correlation coefficient
  Baseline: Heart Rate | 0.01 [-0.43 to 0.44]
  End of Study: Heart Rate | 0.11 [-0.35 to 0.53]
  Baseline: Resting Heart Rate | 0.02 [-0.41 to 0.45]
  End of Study: Resting Heart Rate | 0.1 [-0.36 to 0.52]
  Baseline: Temperature | 0.48 [0.06 to 0.75]
  End of Study: Temperature | 0.21 [-0.25 to 0.6]
  Baseline: Temperature (normalized) | 0.08 [-0.36 to 0.5]
  End of Study: Temperature (normalized) | 0.02 [-0.43 to 0.46]
  Baseline: Respiration Rate | -0.23 [-0.6 to 0.23]
  End of Study: Respiration Rate | -0.14 [-0.55 to 0.32]
  Baseline: SDRR | 0.11 [-0.34 to 0.51]
  End of Study: SDRR | 0.39 [-0.08 to 0.72]
  Baseline: SDNN | 0.17 [-0.29 to 0.56]
  End of Study: SDNN | 0.41 [-0.05 to 0.73]
  Baseline: SDNNI | 0.24 [-0.21 to 0.61]
  End of Study: SDNNI | 0.43 [-0.02 to 0.74]
  Baseline: RMSSD | 0.13 [-0.32 to 0.53]
  End of Study: RMSSD | 0.25 [-0.23 to 0.63]
  Baseline: In (RMSSD) | 0.04 [-0.4 to 0.46]
  End of Study: In (RMSSD) | 0.28 [-0.2 to 0.65]
  Baseline: pNN50 | 0.08 [-0.37 to 0.49]
  End of Study: pNN50 | 0.41 [-0.05 to 0.73]
  Baseline: Stress Index | -0.11 [-0.52 to 0.34]
  End of Study: Stress Index | -0.32 [-0.67 to 0.16]
  Baseline: LF | 0.08 [-0.36 to 0.49]
  End of Study: LF | 0.3 [-0.18 to 0.66]
  Baseline: HF | 0.24 [-0.22 to 0.61]
  End of Study: HF | 0.13 [-0.34 to 0.55]
  Baseline: LF/HF | 0.25 [-0.2 to 0.62]
  End of Study: LF/ HF | 0.16 [-0.32 to 0.57]
  Baseline: Physical Activity | -0.26 [-0.62 to 0.2]
  End of Study: Physical Activity | -0.05 [-0.48 to 0.4]
  Baseline: Physical Activity (normalized) | -0.16 [-0.55 to 0.3]
  End of Study: Physical Activity (normalized) | 0.13 [-0.33 to 0.54]
  Baseline: In- vs. Expiration Time Ratio | -0.34 [-0.68 to 0.1]
  End of Study: In- vs. Expiration Time Ratio | -0.21 [-0.61 to 0.27]
  Baseline: Cough Frequency | -0.53 [-0.78 to -0.13]
  End of Study: Cough Frequency | -0.06 [-0.49 to 0.4]
  Baseline: Cough Frequency (normalized) | 0.24 [-0.21 to 0.61]
  End of Study: Cough Frequency (normalized) | 0.4 [0 to 0.74]

25. Secondary Outcome: Correlation of Sensor-Collected Data With COPD Assessment Test (CAT) Questionnaire: Lung Function and Lab Values at Baseline and Study End (Partial Pressure of Oxygen (pO2))
Description: as for outcome 23
Time Frame: Baseline (Day 0) and at 3 months
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | COPD Cohort
Number analyzed (Participants) | 67
correlation coefficient
  Baseline: Heart Rate | -0.39 [-0.68 to 0.01]
  End of Study: Heart Rate | -0.3 [-0.65 to 0.15]
  Baseline: Resting Heart Rate | -0.41 [-0.69 to -0.01]
  End of Study: Resting Heart Rate | -0.3 [-0.65 to 0.15]
  Baseline: Temperature | -0.3 [-0.62 to 0.11]
  End of Study: Temperature | -0.24 [-0.61 to 0.22]
  Baseline: Temperature (normalized) | 0.02 [-0.38 to 0.41]
  End of Study: Temperature (normalized) | -0.07 [-0.49 to 0.37]
  Baseline: Respiration Rate | -0.54 [-0.77 to -0.19]
  End of Study: Respiration Rate | -0.3 [-0.65 to 0.15]
  Baseline: SDRR | -0.32 [-0.64 to 0.09]
  End of Study: SDRR | -0.27 [-0.64 to 0.21]
  Baseline: SDNN | -0.13 [-0.5 to 0.29]
  End of Study: SDNN | -0.15 [-0.56 to 0.33]
  Baseline: SDNNI | -0.2 [-0.56 to 0.22]
  End of Study: SDNNI | -0.22 [-0.61 to 0.26]
  Baseline: RMSSD | -0.16 [-0.53 to 0.26]
  End of Study: RMSSD | -0.08 [-0.51 to 0.39]
  Baseline: In (RMSSD) | -0.24 [-0.52 to 0.18]
  End of Study: In (RMSSD) | -0.27 [-0.64 to 0.21]
  Baseline: pNN50 | -0.14 [-0.52 to 0.28]
  End of Study: pNN50 | -0.26 [-0.64 to 0.22]
  Baseline: Stress Index | -0.27 [-0.61 to 0.15]
  End of Study: Stress Index | 0.37 [-0.1 to 0.71]
  Baseline: LF | -0.04 [-0.44 to 0.37]
  End of Study: LF | -0.35 [-0.7 to 0.12]
  Baseline: HF | -0.09 [-0.48 to 0.32]
  End of Study: HF | -0.17 [-0.58 to 0.31]
  Baseline: LF/HF | 0.2 [-0.22 to 0.56]
  End of Study: LF/ HF | -0.17 [-0.58 to 0.31]
  Baseline: Physical Activity | 0.47 [0.09 to 0.73]
  End of Study: Physical Activity | -0.05 [-0.47 to 0.39]
  Baseline: Physical Activity (normalized) | 0.24 [-0.18 to 0.58]
  End of Study: Physical Activity (normalized) | -0.17 [-0.56 to 0.28]
  Baseline: In- vs. Expiration Time Ratio | 0.34 [-0.08 to 0.65]
  End of Study: In- vs. Expiration Time Ratio | 0.28 [-0.2 to 0.65]
  Baseline: Cough Frequency | 0.16 [-0.25 to 0.52]
  End of Study: Cough Frequency | 0.24 [-0.21 to 0.61]
  Baseline: Cough Frequency (normalized) | 0.03 [-0.37 to 0.42]
  End of Study: Cough Frequency (normalized) | -0.28 [-0.63 to 0.17]

26. Secondary Outcome: Correlation of Sensor-Collected Data With COPD Assessment Test (CAT) Questionnaire: Lung Function and Lab Values at Baseline and Study End (Partial Pressure of Carbon Dioxide (pCO2))
Description: as for outcome 23
Time Frame: Baseline (Day 0) and at 3 months
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | COPD Cohort
Number analyzed (Participants) | 67
correlation coefficient
  Baseline: Heart Rate | 0.16 [-0.25 to 0.52]
  End of Study: Heart Rate | 0.32 [-0.13 to 0.66]
  Baseline: Resting Heart Rate | 0.18 [-0.23 to 0.54]
  End of Study: Resting Heart Rate | 0.3 [-0.16 to 0.64]
  Baseline: Temperature | 0.13 [-0.28 to 0.5]
  End of Study: Temperature | -0.26 [-0.62 to 0.2]
  Baseline: Temperature (normalized) | 0.54 [0.18 to 0.77]
  End of Study: Temperature (normalized) | -0.55 [-0.8 to -0.16]
  Baseline: Respiration Rate | 0.09 [-0.31 to 0.47]
  End of Study: Respiration Rate | 0.15 [-0.3 to 0.55]
  Baseline: SDRR | -0.04 [-0.43 to 0.37]
  End of Study: SDRR | 0.14 [-0.33 to 0.56]
  Baseline: SDNN | -0.13 [-0.51 to 0.29]
  End of Study: SDNN | -0.12 [-0.55 to 0.35]
  Baseline: SDNNI | -0.16 [-0.53 to 0.26]
  End of Study: SDNNI | -0.04 [-0.49 to 0.42]
  Baseline: RMSSD | -0.14 [-0.51 to 0.28]
  End of Study: RMSSD | -0.32 [-0.67 to 0.16]
  Baseline: In (RMSSD) | -0.21 [-0.56 to 0.21]
  End of Study: In (RMSSD) | -0.29 [-0.66 to 0.19]
  Baseline: pNN50 | -0.14 [-0.52 to 0.28]
  End of Study: pNN50 | -0.14 [-0.56 to 0.34]
  Baseline: Stress Index | 0.45 [0.06 to 0.72]
  End of Study: Stress Index | 0.14 [-0.34 to 0.56]
  Baseline: LF | -0.24 [-0.58 to 0.18]
  End of Study: LF | -0.4 [-0.72 to 0.07]
  Baseline: HF | -0.1 [-0.48 to 0.32]
  End of Study: HF | -0.5 [-0.78 to -0.06]
  Baseline: LF/HF | -0.04 [-0.43 to 0.37]
  End of Study: LF/ HF | 0.23 [-0.25 to 0.62]
  Baseline: Physical Activity | -0.41 [-0.69 to -0.02]
  End of Study: Physical Activity | 0.01 [-0.42 to 0.44]
  Baseline: Physical Activity (normalized) | -0.13 [-0.5 to 0.28]
  End of Study: Physical Activity (normalized) | 0.2 [-0.26 to 0.58]
  Baseline: In- vs. Expiration Time Ratio | -0.3 [-0.63 to 0.11]
  End of Study: In- vs. Expiration Time Ratio | -0.27 [-0.65 to 0.21]
  Baseline: Cough Frequency | -0.27 [-0.6 to 0.14]
  End of Study: Cough Frequency | 0.15 [-0.3 to 0.54]
  Baseline: Cough Frequency (normalized) | 0 [-0.4 to 0.39]
  End of Study: Cough Frequency (normalized) | 0.32 [-0.13 to 0.66]

27. Secondary Outcome: Correlation of Sensor-Collected Data With COPD Assessment Test (CAT) Questionnaire: Lung Function and Lab Values at Baseline and Study End (O2 Saturation)
Description: as for outcome 23
Time Frame: Baseline (Day 0) and at 3 months
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | COPD Cohort
Number analyzed (Participants) | 67
correlation coefficient
  Baseline: Heart Rate | -0.33 [-0.64 to 0.09]
  End of Study: Heart Rate | -0.32 [-0.66 to 0.13]
  Baseline: Resting Heart Rate | -0.35 [-0.66 to 0.06]
  End of Study: Resting Heart Rate | -0.33 [-0.67 to 0.12]
  Baseline: Temperature | -0.29 [-0.62 to 0.13]
  End of Study: Temperature | 0.03 [-0.41 to 0.45]
  Baseline: Temperature (normalized) | -0.28 [-0.61 to 0.14]
  End of Study: Temperature (normalized) | 0.04 [-0.4 to 0.46]
  Baseline: Respiration Rate | -0.28 [-0.61 to 0.14]
  End of Study: Respiration Rate | -0.28 [-0.64 to 0.17]
  Baseline: SDRR | -0.46 [-0.73 to -0.06]
  End of Study: SDRR | -0.37 [-0.7 to 0.11]
  Baseline: SDNN | -0.13 [-0.51 to 0.3]
  End of Study: SDNN | -0.35 [-0.69 to 0.13]
  Baseline: SDNNI | -0.22 [-0.58 to 0.21]
  End of Study: SDNNI | -0.39 [-0.72 to 0.08]
  Baseline: RMSSD | -0.11 [-0.5 to 0.32]
  End of Study: RMSSD | -0.3 [-0.66 to 0.18]
  Baseline: In (RMSSD) | -0.22 [-0.58 to 0.22]
  End of Study: In (RMSSD) | -0.36 [-0.7 to 0.11]
  Baseline: pNN50 | -0.03 [-0.43 to 0.39]
  End of Study: pNN50 | -0.3 [-0.66 to 0.18]
  Baseline: Stress Index | -0.36 [-0.68 to 0.06]
  End of Study: Stress Index | 0.13 [-0.34 to 0.55]
  Baseline: LF | 0.1 [-0.32 to 0.49]
  End of Study: LF | -0.11 [-0.54 to 0.36]
  Baseline: HF | -0.1 [-0.49 to 0.33]
  End of Study: HF | -0.16 [-0.57 to 0.32]
  Baseline: LF/HF | 0.29 [-0.14 to 0.63]
  End of Study: LF/ HF | -0.02 [-0.47 to 0.44]
  Baseline: Physical Activity | 0.44 [0.04 to 0.72]
  End of Study: Physical Activity | 0.1 [-0.34 to 0.51]
  Baseline: Physical Activity (normalized) | 0.17 [-0.25 to 0.53]
  End of Study: Physical Activity (normalized) | -0.07 [-0.48 to 0.38]
  Baseline: In- vs. Expiration Time Ratio | 0.45 [0.04 to 0.73]
  End of Study: In- vs. Expiration Time Ratio | 0.41 [-0.06 to 0.73]
  Baseline: Cough Frequency | 0.04 [-0.37 to 0.44]
  End of Study: Cough Frequency | 0.28 [-0.17 to 0.64]
  Baseline: Cough Frequency (normalized) | -0.11 [-0.5 to 0.3]
  End of Study: Cough Frequency (normalized) | -0.32 [-0.66 to 0.13]

28. Secondary Outcome: Correlation of Sensor-Collected Data With Number, Date of Onset, and Duration of Mild, Moderate, and Severe Exacerbations
Description: Exacerbations are classified as mild if they are treated with short-acting bronchodilators only, moderate if they are treated additionally with antibiotics or oral corticosteroids, or severe if the patient visits the emergency room or requires hospitalization because of an exacerbation.
Time Frame: Up to 3 months
Population: as for outcome 14
Measure: Number; unit: correlation coefficient
Arm/Group | COPD Cohort
Number analyzed (Participants) | 67
correlation coefficient | NA — Data was not evaluable due to low number of exacerbations.

29. Secondary Outcome: Association Between Sensor Parameters (Heart Rate and Resting Heart Rate) and CAT Score
Description: During the observation period the CAT score was obtained via a digital application daily. The daily CAT questionnaire summary score was computed. The fixed effect estimate represents the change in CAT score per unit change in the corresponding parameter. Linear mixed models were performed to assess the association between the CAT score and each sensor parameter (Heart Rate and Resting Heart Rate). Data was calculated through linear mixed model; reported as "fixed effect estimate" with measure type as "number" and measure dispersion as "95% CI."
Time Frame: 7 days before Severe/Moderate Excarbations(S/M E) (7-day window period)
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: scores on a scale/beats per minute
Arm/Group | COPD Cohort
Number analyzed (Participants) | 67
scores on a scale/beats per minute
  7days<S/M E:Heart Rate | 0.039 [0.016 to 0.063]
  7days<S/M E:Resting Heart Rate | 0.039 [0.015 to 0.063]

30. Secondary Outcome: Association Between Sensor Parameters (Respiration Rate) and CAT Score
Description: During the observation period the CAT score was obtained via a digital application daily. The daily CAT questionnaire summary score was computed. The fixed effect estimate represents the change in CAT score per unit change in the corresponding parameter. Linear mixed models were performed to assess the association between the CAT score and each sensor parameter (Respiration Rate). Data was calculated through linear mixed model; reported as "fixed effect estimate" with measure type as "number" and measure dispersion as "95% CI."
Time Frame: 7 days before Severe/Moderate Excarbations(S/M E) (7-day window period) and 14 days before S/M E (1 day window period)
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: scores on a scale/ breaths per minute
Arm/Group | COPD Cohort
Number analyzed (Participants) | 67
scores on a scale/ breaths per minute
  7days<S/M E:Respiration Rate | 0.370 [0.161 to 0.580]
  14days<S/M E:RespirationRate | 0.789 [0.389 to 1.188]

31. Secondary Outcome: Association Between Sensor Parameters (SDRR, SDNN, SDNNI, RMSSD, In(RMSSD)) and CAT Score
Description: During the observation period the CAT score was obtained via a digital application daily. The daily CAT questionnaire summary score was computed. The fixed effect estimate represents the change in CAT score per unit change in the corresponding parameter. Linear mixed models were performed to assess the association between the CAT score and each sensor parameter (SDRR, SDNN, SDNNI, RMSSD, In(RMSSD)). Data was calculated through linear mixed model; reported as "fixed effect estimate" with measure type as "number" and measure dispersion as "95% CI."
Time Frame: 7 days before Severe/Moderate Excarbations(S/M E) (7-day window period) and 14 days before S/M E (1 day window period)
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: scores on a scale/millimeter
Arm/Group | COPD Cohort
Number analyzed (Participants) | 67
scores on a scale/millimeter
  7days<S/M E:SDRR | 0.030 [0.010 to 0.051]
  7days<S/M E:SDNN | 0.010 [0.003 to 0.0171]
  14days<S/M E:SDNN | 0.029 [0.010 to 0.048]
  7days<S/M E:SDNNI | 0.011 [0.003 to 0.018]
  14days<S/M E:SDNNI | 0.045 [0.021 to 0.069]
  7days<S/M E:RMSSD | 0.006 [0.003 to 0.010]
  14days<S/M E:RMSSD | 0.016 [0.004 to 0.027]
  7days<S/M E:In (RMSSD) | 0.576 [0.204 to 0.948]
  14days<S/M E:In(RMSSD) | 1.893 [1.006 to 2.781]

32. Secondary Outcome: Association Between Sensor Parameters (Stress Index, LF/HF) and CAT Score
Description: During the observation period, participants completed the CAT questionnaire daily via a digital app. Stress Index, based on heart rate variability (HRV), assessed autonomic activity and physiological stress. It was calculated as AMo/(2 * Mo * MxDMn), where AMo is the % of RR intervals at the most frequent value, Mo is the most common RR interval, and MxDMn is the RR interval range. Stress Index values range from 50-900; lower values (50-150) indicate low stress and better autonomic balance, while higher values (>500) reflect increased stress and sympathetic activity. LF power reflects sympathetic activity; HF power reflects parasympathetic activity. Linear mixed models assessed associations between CAT score and each sensor parameters. Fixed effect estimates represent change in CAT score per unit change in each parameter. Data was calculated through linear mixed model; reported as "fixed effect estimate" with measure type as "number" and measure dispersion as "95% CI".
Time Frame: 7 days before Severe/Moderate Excarbations(S/M E) (7-day window period) and 14 days before S/M E (1 day window period)
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: fixed effect estimate
Arm/Group | COPD Cohort
Number analyzed (Participants) | 67
fixed effect estimate
  7days<S/M E:Stress Index | 0.003 [0.000 to 0.007]
  14days<S/M E:StressIndex | -0.006 [-0.011 to -0.000]
  7days<S/M E:LF/HF | -0.441 [-0.703 to -0.179]
  14days<S/M E:LF/HF | -0.963 [-1.762 to -0.164]

33. Secondary Outcome: Association Between Sensor Parameters (pNN50) and CAT Score
Description: During the observation period the CAT score was obtained via a digital application daily. The daily CAT questionnaire summary score was computed. The fixed effect estimate represents the change in CAT score per unit change in the corresponding parameter. Linear mixed models were performed to assess the association between the CAT score and each sensor parameter (pNN50). Data was calculated through linear mixed model; reported as "fixed effect estimate" with measure type as "number" and measure dispersion as "95% CI."
Time Frame: 7 days before Severe/Moderate Excarbations(S/M E) (7-day window period) and 14 days before S/M E (1 day window period)
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: scores on a scale/percent of heartbeats
Arm/Group | COPD Cohort
Number analyzed (Participants) | 67
scores on a scale/percent of heartbeats
  7days<S/M E:pNN50 | 2.259 [0.956 to 3.561]
  14days<S/M E:pNN50 | 5.483 [0.723 to 10.242]

34. Secondary Outcome: Association Between Sensor Parameters (Temperature) and CAT Score
Description: During the observation period the CAT score was obtained via a digital application daily. The daily CAT questionnaire summary score was computed. The fixed effect estimate represents the change in CAT score per unit change in the corresponding parameter. Linear mixed models were performed to assess the association between the CAT score and each sensor parameter (Temperature). Data was calculated through linear mixed model; reported as "fixed effect estimate" with measure type as "number" and measure dispersion as "95% CI."
Time Frame: 14 days before S/M E (1 day window period)
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: scores on a scale/degree Celsius
Arm/Group | COPD Cohort
Number analyzed (Participants) | 67
scores on a scale/degree Celsius | 0.943 [0.047 to 1.839]

35. Secondary Outcome: Association Between Sensor Parameters (Physical Activity) and CAT Score
Description: During the observation period the CAT score was obtained via a digital application daily. The daily CAT questionnaire summary score was computed. The fixed effect estimate represents the change in CAT score per unit change in the corresponding parameter. Linear mixed models were performed to assess the association between the CAT score and each sensor parameter (Physical activity). Data was calculated through linear mixed model; reported as "fixed effect estimate" with measure type as "number" and measure dispersion as "95% CI."
Time Frame: 14 days before S/M E (1 day window period)
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: scores on a scale/minute
Arm/Group | COPD Cohort
Number analyzed (Participants) | 67
scores on a scale/minute | -0.016 [-0.031 to -0.000]

36. Secondary Outcome: Association Between Sensor Parameters (Sleep Pattern) and CAT Score
Description: During the observation period the CAT score was obtained via a digital application daily. The daily CAT questionnaire summary score was computed. The fixed effect estimate represents the change in CAT score per unit change in the corresponding parameter. Linear mixed models were performed to assess the association between the CAT score and each sensor parameter (Sleep pattern). Data was calculated through linear mixed model; reported as "fixed effect estimate" with measure type as "number" and measure dispersion as "95% CI."
Time Frame: 14 days before S/M E (1 day window period)
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: scores on a scale/hours per day
Arm/Group | COPD Cohort
Number analyzed (Participants) | 67
scores on a scale/hours per day | -0.292 [-0.571 to -0.014]

37. Secondary Outcome: Predicting the CAT Score by Building a Statistical Model Employing Sensor-Derived Data and Demographic and Medical Covariates
Description: Patients' health status and symptoms at baseline (Day 0) were measured using the CAT questionnaire, an 8-item tool with scores ranging from 0 to 5 per item. CAT scores were collected daily via a digital application during the observation period. Various machine learning algorithms were evaluated for predictive performance using metrics including accuracy, specificity, sensitivity, precision, positive predictive value (PPV), negative predictive value (NPV), and area under the ROC curve. R² (coefficient of determination) was computed for CAT score prediction models, defined as R² = 1 - (SS_res / SS_tot), where SS_res is the residual sum of squares and SS_tot is the total sum of squares. R² values range from 0 to 1, with higher values indicating better model fit.
Time Frame: Up to 3 months
Population: COPD cohort consisted of all participants with COPD fulfilling all of the inclusion criteria and none of the exclusion criteria. Data was not derived due to low number of exacerbations.
Measure: Number; unit: coefficient of determination (R^2)
Arm/Group | COPD Cohort
Number analyzed (Participants) | 67
coefficient of determination (R^2)
  Time-Split Model | 82.7
  XGBoost regressor model | 82.6

ADVERSE EVENTS:
Time Frame: Up to 3 months
Description: No AEs were documented for the calibration cohort and 6 AEs were reported in the COPD cohort
Arm/Group | Calibration Cohort | COPD Cohort
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/67 | 3/67
Other Adverse Events (participants affected / at risk) | 0/67 | 3/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Calibration Cohort (N=67) | COPD Cohort (N=67)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Calibration Cohort (N=67) | COPD Cohort (N=67)
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
The number of moderate or severe exacerbations documented during the observation period was very low.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-03-01): https://cdn.clinicaltrials.gov/large-docs/32/NCT05655832/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/32/NCT05655832/SAP_001.pdf